CLINICAL TRIAL: NCT03121898
Title: PLATelet Function Operating Room Monitoring
Acronym: PLATFORM
Status: Completed | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Marco Ranucci, Head of Cardiothoracic Anesthesia and ICU depy, IRCCS Policlinico S. Donato
Other Study IDs: PlateletMonitoring
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Platelet Dysfunction Due to Drugs; Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — Platelet Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Platelet function test — Measurement of P2Y12 and PAR-dependent platelet function activity before and after cardiac surgery by ADPtest and TRAPtest

SUMMARY:
Prospective cohort study on adult cardiac surgery patients. Platelet function evaluated before and after cardiopulmonary bypass. Bleeding and transfusion recorded. Primary endpoint is finding the association between postoperative platelet function and bleeding.

DETAILED DESCRIPTION:
Preoperative platelet function is a known determinant of postoperative bleeding in cardiac surgery patients (1,2). Conversely, there is a lack of information with respect to postoperative platelet function and postoperative bleeding, and specific cut-off values have not been identified yet.

This study will verify the hypothesis that postoperative platelet function is associated with bleeding, and will test the ability of platelet function tests (PFTs) in predicting severe postoperative bleeding. Additional analyses linking platelet function to other preoperative and intraoperative conditions are planned.

Patients: Enrollment between February 2017 and January 2018. 800 consecutive adult cardiac surgery patients are considered based on our usual surgical activity. Exclusion criteria: unwillingness to participate, known congenital coagulopathy. Moderate/severe bleeding occurs in about 12% of our patient population. Considering a 15% dropout rate, there are about 80 predicted events. Power analysis: to build a predictive model, at least 60 events of moderate/severe bleeding are required. The study will be stopped at reaching (whatever comes first) 800 enrolled pts; 60 events; or 31st January 2018.

Methods: all the patients will receive a preoperative (in the operating room) PFT (ADPtest and TRAPtest) using the aggregometry Multiplate (Roche). The same test will be repeated after protamine administration at the end of CPB.

Definitions of bleeding: 12-hours chest drain blood loss; moderate/severe bleeding adjudicated based on the universal definition of perioperative bleeding (3).

Statistics: ROC analysis with identification of adequate cut-off values and definition of the PPV and NPV

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery with CPB

Exclusion Criteria:

* Known congenital coagulopathy

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cardiac surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Postoperative bleeding | 12 hours
  Chest drain blood loss

SECONDARY OUTCOMES:
Transfusions | 24 hours
  RBC, FFP, and Platelet concentrate transfusions

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ranucci, MD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ranucci M, Baryshnikova E, Soro G, Ballotta A, De Benedetti D, Conti D; Surgical and Clinical Outcome Research (SCORE) Group. Multiple electrode whole-blood aggregometry and bleeding in cardiac surgery patients receiving thienopyridines. Ann Thorac Surg. 2011 Jan;91(1):123-9. doi: 10.1016/j.athoracsur.2010.09.022. PMID 21172499
- [Background] Ranucci M, Colella D, Baryshnikova E, Di Dedda U; Surgical and Clinical Outcome Research (SCORE) Group. Effect of preoperative P2Y12 and thrombin platelet receptor inhibition on bleeding after cardiac surgery. Br J Anaesth. 2014 Dec;113(6):970-6. doi: 10.1093/bja/aeu315. Epub 2014 Sep 10. PMID 25209096
- [Background] Dyke C, Aronson S, Dietrich W, Hofmann A, Karkouti K, Levi M, Murphy GJ, Sellke FW, Shore-Lesserson L, von Heymann C, Ranucci M. Universal definition of perioperative bleeding in adult cardiac surgery. J Thorac Cardiovasc Surg. 2014 May;147(5):1458-1463.e1. doi: 10.1016/j.jtcvs.2013.10.070. Epub 2013 Dec 9. PMID 24332097